CLINICAL TRIAL: NCT05306067
Title: A Prospective Surveillance Study to Detect Antimalarial Drug Resistance, Gene Deletions of Diagnostic Relevance and Genetic Diversity of Plasmodium Falciparum in Mozambique
Brief Title: Plasmodium Falciparum Genomic Intelligence in Mozambique
Acronym: GenMoz
Status: Completed | Type: Observational
Sponsor: Centro de Investigacao em Saude de Manhica (Other)
Collaborators: National Malaria Control Program, Mozambique (Unknown); Malaria Consortium (Other); Barcelona Institute for Global Health (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: GenMoz
Record Dates: First submitted 2022-03-15; First posted 2022-03-31 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Malaria,Falciparum; Malaria in Pregnancy; Malaria
Keywords: drug resistance; diagnostic resistance; surveillance; genomics; importation; genetic diversity; plasmodium falciparum; next generation sequencing; stratification
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Dried blood spot onto filter paper and rapid diagnostic tests collected by finger-prick.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Children at low transmission health facilities
- Children at medium-to-high transmission health facilities
  Interventions: Diagnostic Test: LDH-based malaria rapid diagnostic test
- Pregnant women at low transmission ANC
  Interventions: Diagnostic Test: Malaria rapid diagnostic test
- Pregnant women at medium-to-high transmission transmission ANC
  Interventions: Diagnostic Test: Malaria rapid diagnostic test

INTERVENTIONS:
Diagnostic Test: LDH-based malaria rapid diagnostic test — Malaria testing using an LDH-based malaria rapid diagnostic test will be added to standard routine testing of suspected cases at health facilities
  Groups: Children at medium-to-high transmission health facilities
Diagnostic Test: Malaria rapid diagnostic test — All pregnant women attending their first routine antenatal visit will be tested for malaria using routine malaria rapid diagnostic tests
  Groups: Pregnant women at low transmission ANC; Pregnant women at medium-to-high transmission transmission ANC

SUMMARY:
Mozambique is among the ten countries with the highest burden of malaria worldwide, with an estimated 9.3 million cases in 2018, and constitutes a core target for the World Health Organization (WHO) and the Roll Back Malaria Partnership to End Malaria's country-led 'high burden to high impact' initiative. At the same time, the National Malaria Control Program (NMCP) of Mozambique seeks to accelerate elimination in the south, where transmission is lowest. NMCP is currently working with partners (Malaria Consortium, PMI, Global Fund) to set up a high-resolution surveillance system that can drive decision-making across all transmission strata through strengthening of routine data quality, data use and data to action packages. However, decisions become more complex as control reveals heterogeneity and better tools are required for a strategic use of information to drive impact. The overall objective of the study is to operationalize a functional malaria molecular surveillance (MMS) system that generates reliable and reproducible genomic data over time for programmatic decisions. The integration of genomic data into routine surveillance activities has the potential to increase the actionable intelligence for making programmatic decisions on the optimal mix of control and elimination measures in Mozambique by:

1. Informing drug and diagnostic choices through the monitoring of antimalarial drug resistance and diagnostic resistance (hrp2/3 deletions);
2. Targeting the reservoirs sustaining transmission through the use of transmission network models to quantify parasite importation, identify sources and characterize local transmission in near-elimination settings;
3. Improving stratification, monitoring and impact evaluations in different epidemiological and health system contexts through the use of measures of P. falciparum genetic diversity (routinely from positive cases) to supplement traditional surveillance, especially where it is sparse;
4. Using alternative, cost-effective, approaches targeting easy-access populations (e.g. pregnant women at antenatal care clinics) to monitor transmission and antimalarial/diagnostic resistance.

DETAILED DESCRIPTION:
Genomic data constitutes a valuable adjunct to routine surveillance that can guide programmatic decisions to reduce the burden of infectious diseases. However, genomic capacities remain low in Africa. This study aims to operationalize a functional malaria molecular surveillance system in Mozambique that generates reliable and reproducible genomic data over time for malaria control and elimination. This prospective surveillance study seeks to generate P. falciparum genetic data to 1) monitor molecular markers of drug resistance and deletions in rapid diagnostic test targets; 2) characterize transmission sources (imported/introduced or indigenous) in low transmission settings; and 3) quantify transmission levels and the effectiveness of antimalarial interventions.

Nine provinces were identified through consultation with the NMCP for inclusion in the study: Maputo, Maputo City, Gaza, Inhambane, Niassa, Manica, Nampula, Zambezia and Sofala. Selection of study sites will be stratified by transmission intensity into two major strata: A) low transmission (Maputo province and Maputo City, where individual case notification is in effect for the purpose of a complete interruption of transmission), and B) medium-to-high transmission areas (Gaza, Inhambane, Niassa, Manica, Nampula, Zambezia and Sofala provinces, targeted by control (non-elimination) strategies). The provinces were selected to provide a range of low and medium-to-high transmission intensity, geographies, climatic conditions, malaria interventions mixes and populations (symptomatic, household contacts and sentinel groups). In the low transmission areas, districts and locations will be sampled based on historic surveillance data. Additionally, in Maputo province, the Ponta d'Ouro border post will be included to capture potential imported cases of malaria.

Dried blood spot samples and rapid diagnostic tests will be collected across the study districts through a combination of dense (all malaria cases) and targeted (a selection of malaria cases) sampling of malaria symptomatic cases in low malaria transmission and medium-to-high malaria transmission areas, respectively. In medium-to-high malaria transmission areas a second, non-HRP2 based test will be carried out and discrepant results suggestive of pfhrp2/3 deletions will be recorded and further analysed. Pregnant women attending their first antenatal care visit will be also included to assess their value as sentinel populations for molecular surveillance. Written informed consent will be sought from all survey participants before surveys and blood sample collections are conducted. In that case, information about the purpose of the sample collection will be explained, any questions will be clarified, and written informed consent will be obtained. The information sheet and consent form will also include text explaining informed consent for future use of biological specimens. In case of minors, consent will be sought from parents or guardians. The field worker or nurse will read the informed consent form to adults or the child's parent/guardian and will ask them if he/she agree his/her child to participate in the study. A witness will be required to sign the informed consent in case parent/guardian of the participant is illiterate. The consent will be available in Portuguese and translated into local language spoken at the study areas. The information sheet includes a brief description of the study, the data collection procedure, the blood sample collection procedure, the potential harm to participants, the expected benefits and the voluntary nature of participation at all stages of the interview and blood sampling. Two copies will be signed by the participant and the study team member obtaining the consent. One copy will be given to the participant and the other copy will be kept in the study file at the CISM office.

Sample size per sampling domain has been estimated taking into account antimalarial and diagnostic resistance as a primary use case, considering the negligible carriage of molecular markers of artemisinin resistance and pfhrp2/3 deletions in Mozambique, and setting 5% as the warning threshold. Assuming a 10% of loss of samples or uninterpretable analysis, a sample size of up to 500 per sampling domain would be adequate to: a) estimate a proportion of 0.05 (markers of drug resistance or pfhrp2 deletion) with 0.026 absolute precision and 95% confidence and b) achieve a power of 80% for detecting an increase of genetic marker (resistance or deletion) from 0 ‰ to 5% at a two-sided p-value of 0.01. It is estimated that up to 500 participants will be recruited among all ages for the study in each sampling unit (i.e. province) across those accessing APEs and health facilities (except Maputo city and Maputo province where continuous collections may exceed this number and household contact sample collection may increase this further). We will target up 500 RDT-positive pregnant women attending ANC clinics in all medium-to-high transmission districts and in low transmission areas each year for a period of three years. A flexible and adaptive sampling scheme will be followed, where a) estimates generated during the first half of the project will inform subsequent sampling schemes and b) not all the samples collected will be analysed (some of them will be stored as reference materials or for confirmation of findings).

The project will also leverage from intervention studies and surveillance activities being conducted in Mozambique between 2021 and 2024, namely: the Malaria Indicator Survey (2022-2023) in southern Mozambique; the Therapeutic Efficacy Survey (2022) in sentinel sites in the country (Cabo Delgado, Tete, Sofala, Zambézia and Inhambane); reactive surveillance activities (Maputo province); a Phase III cluster-randomized, open-label, clinical trial to study the safety and efficacy of ivermectin mass drug administration to reduce malaria transmission (Zambezia; 2022); a large-scale implementation development project aiming at maximising the delivery and uptake of intermittent preventive treatment in infancy (IPTi) (Inhambane; 2022-2024); a hybrid effectiveness-implementation study to evaluate the feasibility and effectiveness of seasonal malaria chemoprevention (SMC) with sulfadoxine-pyrimethamine and amodiaquine (Nampula; 2022); and a programmatic delivery of a population-based mass drug administration with dihydroartemisinin-piperaquine (Gaza Province; 2022-2023).

Molecular analysis will be conducted at CISM. Initial planned genomic analyses of parasite DNA are as follows, though it is possible that improved technologies, protocols, and/or additional parasite genomic targets of interest may become apparent during the course of this project, in part from lessons learned from the data generated herein. Informative SNPs and short haplotypes will be targeted using multiplexed primers on flanking sequences, with a range of amplicon size of ~150-250 bp (covered by a paired end read). Targeted amplicons obtained by PCR on genomic DNA using universal tags, Illumina-specific adaptors and sample-specific barcode will be pooled to create a single product library, which will be sequenced (paired-end 150-bp) on an Illumina MiSeq or NextSeq. Alternative molecular approaches will be used if the single multiplexed amplicon approach does not provide the expected results. Samples will be also used for other molecular analysis of programmatic interest, such as the detection of Plasmodium species, parasite antigens, serological markers of parasite exposure (antibodies)and parasite RNA-based markers (i.e., gametocytes). For quality control purposes, up to 5% of the analysed samples will be transported to UCSF (USA) and/or ISGlobal (Spain) for secondary analysis.

Sequences generated through the analysis of samples collected (from Mozambique and neighbouring countries) will be integrated into a curated catalogue of genomic data together with relevant clinical and epidemiological information. These databases will be made publicly available in open access repositories such as the European Nucleotide Archive (ENA) and MalariaGen Resource Center. In order to facilitate data accessibility and use, and to obtain a meaningful integration with other sources of surveillance data, genetic information will be incorporated into the DHIS2-based Integrated malaria information storage system (iMISS), which is currently being rolled out. The iMISS includes: case data, focus investigations, entomological surveillance data and intervention data. Data visualizations, and dashboards will be defined in collaboration with all users and stakeholders and aligned with the current work led by WHO GMP regarding standardization of malaria dashboards. We will establish risk profile algorithms and interpretation components that are capable of generating outputs on a) country-wide antimalarial resistance profiles (rolling-basis); b) in very low transmission areas, genetic connectivity and case classification (together with travel history and other parameters obtained from case-based notification tools); and c) "high burden to high impact"-specific analysis (i.e., stratification and trend analyses for exploring the potential impact of intervention mixes implemented), to be agreed in consultation with WHO and the SM&E TWG.

ELIGIBILITY:
A) LOW TRANSMISSION AREAS

Inclusion Criteria:

* Any age
* Fever (axillary temperature ≥37.5ºC) or history of fever in the preceding 24 hours
* Positive parasitological test for malaria diagnosis via RDT or microscopy OR
* Household contact of someone with fever/history of fever and Pf positive RDT
* Positive parasitological test for malaria diagnosis via RDT OR
* Pregnant women attending first antenatal care visit AND
* Informed, written consent to participate from participant and/or guardian

Exclusion Criteria:

* Any symptoms of severe malaria
* Negative parasitological test for malaria via RDT or microscopy (except any women at their first ANC visit, who will be recruited before testing for malaria with an RDT)
* Unwilling to provide informed, written consent
* History of antimalarial treatment in the last 14 days

B) MEDIUM-TO-HIGH TRANSMISSION AREAS

Inclusion Criteria:

* Children 2-10 years of age
* Fever (axillary temperature ≥37.5ºC) or history of fever in the preceding 24 hours
* Positive parasitological test for malaria diagnosis via RDT or microscopy OR
* Pregnant women attending first antenatal care visit AND
* Informed, written consent to participate from participant and/or guardian

Exclusion Criteria:

* Any symptoms of severe malaria
* Negative parasitological test for malaria via RDT or microscopy (except any women at their first ANC visit, who will be recruited before testing for malaria with an RDT)
* Unwilling to provide informed, written consent
* History of antimalarial treatment in the last 14 days

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: In low transmission areas, people of any age (> 6 months of age), with clinical symptoms of malaria and a parasitologically confirmed malaria diagnosis via RDT or microscopy will be invited to participate in the study, along with any household contacts of these malaria index cases, if they test P. falciparum positive with an RDT. Malaria-positive index cases of all ages from Magude and Matutuine will be also recruited, as well as individuals crossing the Matutuine Ponta d'Ouro border post who have a malaria positive RDT. In medium-to-high transmission areas, children under 2-10 years old, with clinical symptoms of malaria and a P. falciparum positive RDT will be invited to participate. Pregnant women attending their first antenatal care visit (any trimester) will be invited to participate in both trasnmission areas.
Sampling Method: Non-Probability Sample
Enrollment: 21848 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of molecular markers of diagnostic resistance and antimalarial drug resistance by period, study area and population | Year 3
Genetic diversity of the parasite population by period, study area and population | Year 3
Genetic relatedness between pairs of samples and populations by period, study area and population | Year 3

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Investigaçao em Saúde de Manhiça, Manhiça, Maputo Province, Mozambique

REFERENCES:
- [Derived] Mayor A, da Silva C, Rovira-Vallbona E, Roca-Feltrer A, Bonnington C, Wharton-Smith A, Greenhouse B, Bever C, Chidimatembue A, Guinovart C, Proctor JL, Rodrigues M, Canana N, Arnaldo P, Boene S, Aide P, Enosse S, Saute F, Candrinho B. Prospective surveillance study to detect antimalarial drug resistance, gene deletions of diagnostic relevance and genetic diversity of Plasmodium falciparum in Mozambique: protocol. BMJ Open. 2022 Jul 12;12(7):e063456. doi: 10.1136/bmjopen-2022-063456. PMID 35820756
- See also: MESA Track project registration — https://mesamalaria.org/mesa-track/genmoz-plasmodium-falciparum-genomic-intelligence-mozambique